CLINICAL TRIAL: NCT03871556
Title: Diagnostic Ultrasound for Measuring Fat of the Body
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Murad Alam, Principal Investigator, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STU002089391
Record Dates: First submitted 2019-02-12; First posted 2019-03-12 (Actual); Results first posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Subcutaneous Fat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Experimental Group (Experimental)
  Interventions: Diagnostic Test: LOGIQ P6 Diagnostic Ultrasound

INTERVENTIONS:
Diagnostic Test: LOGIQ P6 Diagnostic Ultrasound — Ultrasound measurements of subcutaneous fat thickness

SUMMARY:
The purpose of this study is to provide information about human subcutaneous fat thickness at different anatomic sites on the body by measuring these thicknesses with a diagnostic ultrasound and also by correlating patient perceptions of body image with measured fat distribution.

Subjects currently living in the Chicago metropolitan area and meet inclusion/exclusion criteria will be considered for enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Males or females 18-85 years old.
* Subjects are in good health as judged by the investigator.
* Subjects with Body Mass Index (BMI) between 18-29.99.
* Subjects who are willing and have the ability to understand and provide informed consent for participation in the study and are able to communicate with the investigator

Exclusion Criteria:

* Evidence of another skin condition affecting the treatment area that would interfere with clinical assessments
* Pregnant or breast feeding
* Uncooperative patients or patients with neurological disorders who are incapable of following directions
* Subjects who are unable to understand the protocol or give informed consent (including non-English speaking patients)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2022-10-02 (Actual); Study Completion 2022-10-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Murad Alam, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Department of Dermatology, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Experimental Group
Started | 40
Completed | 40
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Experimental Group
Number analyzed (Participants) | 40
Age, Customized [Count of Participants; unit: Participants]
  Age: 20-30 | 15
  Age: 31-40 | 8
  Age: 41-50 | 6
  Age: 51-60 | 7
  Age: 61-70 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 8
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 18
  More than one race | 4
  Unknown or Not Reported | 0
Education [Count of Participants; unit: Participants]
  Some high school or less | 0
  High school diploma/GED | 3
  Vocational school or some college, including 2 years degree | 14
  4-year college degree | 11
  Professional or graduate degree | 12
Job status [Count of Participants; unit: Participants]
  Full time | 35
  Part time | 1
  Self-employed | 1
  Unemployed | 0
  Retired | 1
  Homemaker | 0
  Other | 2
Body Mass Index (BMI) [Count of Participants; unit: Participants]
  Less than 18.5 | 0
  18.5-24.9 | 12
  25.0-29.9 | 15
  30 or higher | 13

OUTCOME MEASURES:

1. Primary Outcome: Difference in Thickness of Subcutaneous Fat at Different Anatomic Sites on the Body
Description: Will use diagnostic ultrasound to measure fat thickness
Time Frame: through study completion, 1 day
Measure: Mean (Standard Deviation); unit: average fat measurement (cm)
Groups:
- Male; Female: LOGIQ P6 Diagnostic Ultrasound: Ultrasound measurements of subcutaneous fat thickness
Arm/Group | Male | Female
Number analyzed (Participants) | 18 | 22
average fat measurement (cm)
  Chin | .56 (.27) | .60 (.14)
  Left arm | .83 (.59) | 1.65 (.57)
  Right arm | .82 (.51) | 1.72 (.58)
  Left back | .77 (.44) | 1.30 (.45)
  Right back | .86 (.51) | 1.20 (.52)
  Left flank | 1.31 (.58) | 1.81 (.47)
  Right flank | 1.16 (.55) | 1.83 (.47)
  Abdomen | 1.71 (.70) | 2.19 (.61)
  Left inner thigh | .86 (.58) | 1.40 (.57)
  Right inner thigh | .88 (.63) | 1.41 (.57)
  Left outer thigh | 1.47 (.63) | 2.45 (1.56)
  Right outer thigh | 1.19 (.63) | 2.22 (.57)

2. Primary Outcome: Gender Differences on Patient Perceptions of Body Image With Measured Fat Distribution
Description: Will use diagnostic ultrasound to measure fat thickness and a questionnaire to assess subject perceptions of their body using a 10-point Likert scale (1= very unsatisfied, 10= very satisfied)
Time Frame: through study completion, 1 day
Measure: Mean (Standard Deviation); unit: average satisfaction level
Arm/Group | Male | Female
Number analyzed (Participants) | 18 | 22
average satisfaction level
  Chin | 8.48 (1.38) | 5.14 (3.47)
  Inner arms | 7.41 (2.45) | 4.02 (3.22)
  Upper back | 7.90 (1.91) | 5.18 (2.81)
  Flanks | 6.48 (2.6) | 3.45 (2.97)
  Abdomen | 5.98 (2.71) | 2.93 (3.12)
  Inner thigh | 7.58 (2.12) | 5.04 (3.62)
  Outer thigh | 7.91 (2.25) | 5.93 (3.15)
  Overall | 7.28 (2.13) | 4.70 (2.24)

ADVERSE EVENTS:
Time Frame: One 3 hour session on 1 day
Arm/Group | Experimental Group
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-10-10): https://cdn.clinicaltrials.gov/large-docs/56/NCT03871556/Prot_SAP_000.pdf
  • Informed Consent Form (2018-10-10): https://cdn.clinicaltrials.gov/large-docs/56/NCT03871556/ICF_001.pdf